CLINICAL TRIAL: NCT02551094
Title: Colchicine Cardiovascular Outcomes Trial (COLCOT)
Acronym: COLCOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MHIPS-003
Record Dates: First submitted 2015-08-26; First posted 2015-09-16 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colchicine (Active Comparator): 0.5 mg tablet of colchicine taken once a day
  Interventions: Drug: colchicine
- colchicine placebo (Placebo Comparator): 0.5 mg tablet of placebo taken once a day
  Interventions: Drug: colchicine placebo

INTERVENTIONS:
Drug: colchicine — 0.5 mg tablet taken once a day
  Other Names: no other name
  Arms: colchicine
Drug: colchicine placebo — sugar pill manufactured to mimic colchicine 0.5 mg tablet
  Other Names: no other name
  Arms: colchicine placebo

SUMMARY:
The study evaluates whether long-term treatment with colchicine reduces rates of cardiovascular events in patients after myocardial infarction. Patients who have suffered a documented acute myocardial infarction within the last 30 days, are treated according to the national guidelines and after having completed any planned percutaneous revascularization procedures associated with their initial infarction will receive either colchicine (0.5 mg per day) or matching placebo (1:1 allocation ratio) for an estimated 2 years period or until the target of 301 primary endpoints has been reached.

DETAILED DESCRIPTION:
Atherosclerosis is the most common cause of myocardial infarction, stroke and peripheral arterial disease. Research has clearly demonstrated that inflammation plays a key role in the initiation, progression and manifestations of atherosclerosis. Atherosclerotic lesions begin as an accumulation of lipid-laden cells (primarily macrophages) beneath the endothelium, and progress with the further accumulation of cells, connective-tissue elements, lipids and debris through immunological and inflammatory activation. Neutrophils and other inflammatory cells have been shown to invade culprit atherosclerotic lesions in acute coronary syndromes. It is likely that the inflammatory process is responsible for the high rate of cardiovascular events despite significant advances in the treatment of risk factors such as hypercholesterolemia and hypertension. It is vital to improve our understanding of the inflammatory nature of atherosclerotic disease and modify the inflammatory process with targeted therapies. Prospective cohort studies have consistently shown that high sensitivity C-reactive protein (hs-CRP) and several other biomarkers of inflammation are independently associated with increasing risk of future cardiovascular events in different populations. This together with animal models showing that reduced inflammation has anti-atherosclerotic effects, create the impetus to test the hypothesis that treatment of the underlying inflammatory process will contribute to improved cardiovascular clinical outcomes. Colchicine is an inexpensive, yet potent, anti-inflammatory drug approved for acute use in patients with gout and chronic use in patients with Familial Mediterranean Fever. The mechanism of action is through the inhibition of tubulin polymerization and potentially also through effects on cellular adhesion molecules and inflammatory chemokines. Colchicine may also have direct anti-inflammatory effects by inhibiting key inflammatory signaling networks known as the inflammasome and pro-inflammatory cytokines. Through the disruption of the cytoskeleton, colchicine is believed to suppress secretion of cytokines and chemokines as well as in vitro platelet aggregation. Considerable work has highlighted the potential of colchicine in the treatment of cardiovascular diseases mediated by pro-inflammatory processes. More recently colchicine has been evaluated for its effect on cardiovascular events in patients with coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* Males and females of at least 18 years of age capable and willing to provide informed consent
* Patient must have suffered a documented acute myocardial infarction within the last 30 days
* Patient must be treated according to national guidelines (including anti-platelet therapy, statin, renin-angiotensin-aldosterone system inhibitor (preferably angiotensin-converting enzyme) and beta-blocker when indicated)
* Patient must have completed any planned percutaneous revascularization procedures associated with his or her qualifying myocardial infarction
* Female patient is either not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile, or is of childbearing potential and practicing at least one method of contraception and preferably two complementary forms of contraception
* Patient is judged to be in good general health as determined by the principal investigator
* Patient must be able and willing to comply with the requirements of this study protocol

Exclusion Criteria:

* Patient with a poorly controlled medical condition, such as New York Heart Association Class III-IV heart failure, a left ventricular ejection fraction of less than 35%, recent stroke (within the past 3 months), or any other condition which in the opinion of the investigator, would put the patient at risk if participating in this study
* Patient with a Type 2 index MI (secondary to ischemic imbalance)
* Patient with a prior coronary artery bypass graft within the past 3 years, or planned
* Patient currently in cardiogenic shock or with hemodynamic instability
* Patient with a history of cancer or lymphoproliferative disease within the last 3 years other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and or localized carcinoma in situ of the cervix
* Patient with inflammatory bowel disease (Crohn's disease or ulcerative colitis) or patient with chronic diarrhea
* Patient with pre-existent progressive neuromuscular disease or patient with creatine phosphokinase level greater than 3 times the upper limit of normal (unless due to myocardial infarction which is allowed) as measured within the past 30 days and determined to be non-transient through repeat testing
* Patient with any of the following as measured within the past 30 days, and determined to be non-transient through repeat testing: hemoglobin less than 115 grams/L, white blood cell count less than 3.0 X 10(9)/L,platelet count less than 110 X 10(9)/L, alanine aminotransferase greater than 3 times the upper limit of normal, total bilirubin greater than 2 times the upper limit of normal (unless due to Gilbert syndrome, which is allowed), creatinine greater than 2 times the upper limit of normal
* Patient with a history of cirrhosis, chronic active hepatitis or sever hepatic disease
* Female patient who is pregnant, or breast-feeding or is considering becoming pregnant during the study or for 6 months after the last dose of study medication
* Patient with a history of clinically significant drug or alcohol abuse in the last year
* Patient is currently using or plan to begin chronic systemic steroid therapy (oral or intravenous) during the study (topical or inhaled steroids are allowed)
* Patient currently taking colchicine for other indications (mainly chronic indications represented by Familial Mediterranean Fever or gout); there is no wash-out period required for patients who have been treated with colchicine and stopped treatment prior to enrollment
* Patient with history of an allergic reaction or significant sensitivity to colchicine
* Patient who has used an investigational chemical agent less than 30 days or 5 half-lives prior to the screening visit (whichever is longer)
* Patient is considered by he investigator, for any reason, to be an unsuitable candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4745 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute; Andreas Orfanos, MD, Study Director — Montreal Health Innovations Coordinating Centre
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bouabdallaoui N, Tardif JC, Waters DD, Pinto FJ, Maggioni AP, Diaz R, Berry C, Koenig W, Lopez-Sendon J, Gamra H, Kiwan GS, Blondeau L, Orfanos A, Ibrahim R, Gregoire JC, Dube MP, Samuel M, Morel O, Lim P, Bertrand OF, Kouz S, Guertin MC, L'Allier PL, Roubille F. Time-to-treatment initiation of colchicine and cardiovascular outcomes after myocardial infarction in the Colchicine Cardiovascular Outcomes Trial (COLCOT). Eur Heart J. 2020 Nov 7;41(42):4092-4099. doi: 10.1093/eurheartj/ehaa659. PMID 32860034
- [Derived] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colchicine | Colchicine Placebo
Started | 2366 | 2379
Completed | 2226 | 2232
Not Completed | 140 | 147

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | Colchicine Placebo | Total
Number analyzed (Participants) | 2366 | 2379 | 4745
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.7) | 60.5 (10.6) | 60.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 472 | 437 | 909
  Male | 1894 | 1942 | 3836
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: Asian | 26 | 27 | 53
  Ethnic Origin: Asian and Caucasian | 1 | 1 | 2
  Ethnic Origin: Black or African American | 3 | 8 | 11
  Ethnic Origin: Black or African American and Caucasian | 1 | 0 | 1
  Ethnic Origin: Black or African American and Hispanic or Latino | 1 | 1 | 2
  Ethnic Origin: Caucasion | 1350 | 1329 | 2679
  Ethnic Origin: Caucasian and Hispanic or Latino | 17 | 18 | 35
  Ethnic Origin: Hispanic or Latino | 377 | 381 | 758
  Ethnic Origin: Indian ancestry | 1 | 0 | 1
  Ethnic Origin: Metis, aboriginal | 0 | 1 | 1
  Ethnic Origin: Native American | 3 | 5 | 8
  Ethnic Origin: North African / Middle Eastern | 70 | 73 | 143
  Ethnic Origin: France n=1051 (Ethnic origin was not provided | 516 | 535 | 1051
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 230 | 226 | 456
  Canada | 739 | 744 | 1483
  Chile | 111 | 108 | 219
  Colombia | 82 | 84 | 166
  France | 516 | 535 | 1051
  Germany | 6 | 2 | 8
  Italy | 270 | 260 | 530
  Lebanon | 92 | 88 | 180
  Portugal | 111 | 116 | 227
  Spain | 32 | 31 | 63
  Tunisia | 100 | 100 | 200
  United Kingdom | 77 | 77 | 154

OUTCOME MEASURES:

1. Primary Outcome: First Event of Cardiovascular Death, Resuscitated Cardiac Arrest, Acute Myocardial Infarction, Stroke, or Urgent Hospitalization for Angina Requiring Coronary Revascularization
Description: The descriptive statistics are the number of participants having at least one of the composites of the primary endpoint.
Time Frame: From randomization to occurence of first event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 170 | 131

2. Secondary Outcome: Death (Total Mortality)
Description: The descriptive statistics are the number of participants having deceased.
Time Frame: From randomization to death, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 44 | 43

3. Secondary Outcome: Cardiovascular Death
Description: The descriptive statistics are presented as the number of participants having had a cardiovascular death.
Time Frame: From randomization to death, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 24 | 20

4. Secondary Outcome: Resuscitated Cardiac Arrest
Description: The descriptive statistics are presented as the number of participants having had resuscitated cardiac arrest
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 6 | 5

5. Secondary Outcome: Myocardial Infarction
Description: The descriptive statistics are presented as the number of participants having had myocardial infarction.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 98 | 89

6. Secondary Outcome: Stroke
Description: The descriptive statistics are presented as the number of participants having had a stroke.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 19 | 5

7. Secondary Outcome: Urgent Hospitalization for Angina Requiring Coronary Revascularization
Description: The descriptive statistics are presented as the number of participants having had urgent hospitalization for angina requiring coronary revascularization.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 50 | 25

8. Secondary Outcome: First Event of Cardiovascular Death, Resuscitated Cardiac Arrest, Acute MI or Stroke.
Description: The descriptive statistics are presented as the number of participants having had a first event of cardiovascular death, resuscitated cardiac arrest, acute MI or stroke.
Time Frame: From randomization to occurence of first event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 130 | 111

9. Other Pre Specified Outcome: First Event of Deep Venous Thrombosis or Pulmonary Embolus
Description: The descriptive statistics are presented as the number of participants having had a first event of deep venous thrombosis or pulmonary embolus.
Time Frame: From randomization to occurence of first event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 7 | 10

10. Other Pre Specified Outcome: Atrial Fibrillation
Description: The descriptive statistics are presented as the number of participants having had atrial fibrillation.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 40 | 36

11. Other Pre Specified Outcome: Heart Failure Hospitalization
Description: The descriptive statistics are presented as the number of participants having had heart failure hospitalization.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 18 | 25

12. Other Pre Specified Outcome: Coronary Revascularization
Description: The descriptive statistics are presented as the number of participants having had coronary revascularization.
Time Frame: From randomization to event, assessed up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine Placebo | Colchicine
Number analyzed (Participants) | 2379 | 2366
Participants | 164 | 132

ADVERSE EVENTS:
Time Frame: The time period covered was from randomization to last follow up which lasted 3.5 years.
Arm/Group | Colchicine Placebo | Colchicine
All-Cause Mortality (participants affected / at risk) | 44/2346 | 41/2330
Serious Adverse Events (participants affected / at risk) | 404/2346 | 383/2330
Other Adverse Events (participants affected / at risk) | 371/2346 | 372/2330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Placebo (N=2346) | Colchicine (N=2330)
Gastro-intestinal SAE (Gastrointestinal disorders) | 36 (404) | 46 (383)
Infection SAE (Infections and infestations) | 38 (404) | 51 (383)
Pneumonia SAE (Respiratory, thoracic and mediastinal disorders) | 9 (404) | 21 (383)
Septic Shock SAE (Infections and infestations) | 2 (404) | 2 (383)
Other (General disorders) | 319 (404) | 263 (383)
HF hospitalization SAE (Cardiac disorders) | 17 (371) | 25 (383)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Placebo (N=2346) | Colchicine (N=2330)
Diarrhea AE (Metabolism and nutrition disorders) | 208 (371) | 225 (372)
Nauseau AE (Gastrointestinal disorders) | 24 (371) | 43 (372)
Flatulence AE (Gastrointestinal disorders) | 5 (371) | 15 (372)
GI Haemorrhage AE (Gastrointestinal disorders) | 5 (371) | 7 (372)
Anaemia AE (Blood and lymphatic system disorders) | 10 (371) | 14 (372)
Leukopenia AE (Blood and lymphatic system disorders) | 3 (371) | 2 (372)
Thrombocytopenia AE (Blood and lymphatic system disorders) | 7 (371) | 3 (372)
Other (General disorders) | 109 (371) | 63 (372)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02551094/SAP_000.pdf
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT02551094/Prot_001.pdf